CLINICAL TRIAL: NCT03033030
Title: Tomosynthesis (TS) or Ultrasound (US) in Mammography-negative Dense Breasts (TOMUS). National Multicenter Trial
Acronym: TOMUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Genova (Other)
Responsible Party: Principal Investigator, Alberto Tagliafico, Assistant Professor, University of Genova
Other Study IDs: 102REG2016
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Breast Cancer
Keywords: Ultrasound; Digital Breast Tomosynthesis; Cancer Detection rate; Sensitivity; Specificity; Breast density
MeSH Terms: conditions — Breast Neoplasms; Hypersensitivity | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tomosynthesis: Patients undergoing Digital Breast Tomosynthesis
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Ultrasound examination

SUMMARY:
Breast cancer remains a worldwide big killer with a rate of deaths compared with newly diagnosed cases not lower than 20%. Mammography is the primary imaging modality for the early detection of clinically occult breast cancer. Mammography is established as the primary investigation for population-based breast cancer screening. Advances in mammographic technique regarding both hardware and software applications are still not sufficient to overcome mammography's limitation with regard to both sensitivity and specificity. Depending on several factors, such as age and breast density, mammography screening is associated with a false-negative rate of 10-20 %.

Digital Breast Tomosynthesis (TS) is a novel technique that is able to study the breast using 3D reconstructions of the tissue from multiple low-dose digital mammographic images acquired in several planes in a 15 to 50 degree angle. This process aims at a increasing the number of lesion visible due to the reduction of overlapping breast tissue.

In TS, to overcome these limitations, a digital mammography (DM) unit is modified to allow the X-ray tube to move through a proscribed arc of excursion acquiring a fixed number of discrete projection images while the breast remains in compression. The individual projection images are extremely low in dose, so the composite dose incurred during a TS acquisition may be similar to that of a standard 2D mammography. The radiologically dense breasts are associated with decreased sensitivity of mammography, both in the clinical and screening setting as well as its established association with breast cancer risk. The systematic application of ultrasound (US) in women with radiologically dense breasts and negative mammogram has been shown to be associated with an additional cancer detection rate [7,8,9]. Incremental ultrasound detection of cancer may be considered in the range of 0.27% to 0.52% of ultrasound-screened women in different density categories [10]. In addition, the main limitation of US in breast screening is represented by false- positive findings. These findings result in additional investigation or unnecessary surgical biopsy [10].

DETAILED DESCRIPTION:
Breast cancer remains a worldwide big killer with a rate of deaths compared with newly diagnosed cases not lower than 20%. Mammography is the primary imaging modality for the early detection of clinically occult breast cancer. Mammography is established as the primary investigation for population-based breast cancer screening. Advances in mammographic technique regarding both hardware and software applications are still not sufficient to overcome mammography's limitation with regard to both sensitivity and specificity. Depending on several factors, such as age and breast density, mammography screening is associated with a false-negative rate of 10-20 %.

Digital Breast Tomosynthesis (TS) is a novel technique that is able to study the breast using 3D reconstructions of the tissue from multiple low-dose digital mammographic images acquired in several planes in a 15 to 50 degree angle. This process aims at a increasing the number of lesion visible due to the reduction of overlapping breast tissue.

In TS, to overcome these limitations, a digital mammography (DM) unit is modified to allow the X-ray tube to move through a proscribed arc of excursion acquiring a fixed number of discrete projection images while the breast remains in compression. The individual projection images are extremely low in dose, so the composite dose incurred during a TS acquisition may be similar to that of a standard 2D mammography. The radiologically dense breasts are associated with decreased sensitivity of mammography, both in the clinical and screening setting as well as its established association with breast cancer risk. The systematic application of ultrasound (US) in women with radiologically dense breasts and negative mammogram has been shown to be associated with an additional cancer detection rate. Incremental ultrasound detection of cancer may be considered in the range of 0.27% to 0.52% of ultrasound-screened women in different density categories [10]. In addition, the main limitation of US in breast screening is represented by false- positive findings. These findings result in additional investigation or unnecessary surgical biopsy.

The study aims to demonstrate at least statistical equivalence, or non-significant difference between TS and US in women with dense breasts.

If the equivalence between TS and US will be demonstrated, US may be substituted by TS with great benefits for the patients and for the healthcare resources we aim to:

1. Assess if TS may detect additional cancers in dense breasts that approximate US detection capability but with less false positive findings than US.
2. If TS detects new cancers in dense breasts similarly to US (approximate rate or marginally lower rate), evaluate the true positive/false positive ratio.
3. Cost-analysis. In case of less false positives detected by TS, the TP/ FP trade-off might be strongly in favour of TS with a great potential of costs reduction.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic subjects <50 years of age presenting for mammography, with the exception of those that, on previous mammograms are found to have breast density BI- RADS D1-2.
* Asymptomatic subjects ≥ 50 years of age who request mammography and have breast density BI-RADS 3-4.
* Written Informed consent.

Exclusion Criteria:

* Pregnant and breast feeding women
* Unable to tolerate breast compression
* Breast implants
* Unable to understand or execute written informed consent
* Unable or unwilling to agree to follow-up during observation period

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who undergo breast TS and Mammography
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2014-02 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Incremental Cancer Detection Rate or Area Under the Curve | 2 years
  The study aims to demonstrate at least statistical equivalence, or non-significant difference between TS and US in women with dense breasts.

SECONDARY OUTCOMES:
TP/FP rate | 2 years
  If the equivalence between TS and US will be demonstrated, US may be substituted by TS with great benefits for the patients and for the healthcare resources we aim to:
  1. Assess if TS may detect additional cancers in dense breasts that approximate US detection capability but with less false positive findings than US.
  2. If TS detects new cancers in dense breasts similarly to US (approximate rate or marginally lower rate), evaluate the true positive/false positive ratio.
  3. Cost-analysis. In case of less false positives detected by TS, the TP/ FP trade-off might be strongly in favour of TS with a great potential of costs reduction.

CONTACTS AND LOCATIONS:
Locations (1):
- UNIGE, Genova, Genova, Italy